CLINICAL TRIAL: NCT03277547
Title: The Association of Biomarkers of Endothelial Function With Prospective Changes in Kidney Function in Sickle Cell Anemia
Brief Title: Kidney Function in Sickle Cell Anemia
Status: Active, not recruiting | Type: Observational
Sponsor: Kenneth Ataga MD (Other)
Collaborators: Ohio State University (Other); University of North Carolina (Other)
Responsible Party: Sponsor-Investigator, Kenneth Ataga MD, Professor, University of Tennessee
Organization: University of Tennessee (Other)
Other Study IDs: 17-0936; 1R01FD006030-01 (FDA)
Record Dates: First submitted 2017-09-01; First posted 2017-09-11 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Sickle Cell Disease; Kidney Failure, Chronic
MeSH Terms: conditions — Anemia, Sickle Cell; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples will be collected to measure biomarkers of endothelial function. Plasma and urine samples will be collected for measurement of metabolic profiles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective clinical cohort study that involves a baseline study visit followed by up to 3 annual follow-up study visits for a total follow-up of 36-48 months to evaluate the age- and sex-adjusted rate of change in kidney function, and to identify biomarkers of endothelial function, metabolomic profiles and clinical characteristics for the worsening of kidney function and for a rapid decline in kidney function.

"Funding Source - FDA OOPD"

DETAILED DESCRIPTION:
Sickle cell disease is a severe monogenic disorder which affects approximately 80,000 patients in the US. It is characterized by a vasculopathy with involvement of multiple organs and resulting in complications such as ischemic stroke, pulmonary hypertension, autosplenectomy, priapism, as well as chronic kidney disease (CKD). Despite the high prevalence of CKD and its known association with increased mortality, the natural history of CKD and the factors associated with changes in kidney function in patients with SCD remain incompletely defined. Furthermore, the available treatment options for albuminuria, an early manifestation of CKD, in patients with SCD are limited. In fact, no controlled studies have confirmed the long-term efficacy of angiotensin-converting enzyme (ACE) inhibitors, the current "standard of care." There is increasing evidence for a contribution of endothelial dysfunction to the pathophysiology of albuminuria in SCD. The association of biomarkers of endothelial function with albuminuria provides opportunities, not only to assess the effect of therapies which improve endothelial function, but also to evaluate the predictive value of these biomarkers for a decline in kidney function. The long-range goal is to develop a model to identify patients at particularly high risk for a decline in kidney function.

In this study, the investigators will evaluate rate of change in kidney function (decline in estimated glomerular filtration rates and increase in albuminuria) and identify biomarkers of endothelial function, metabolomic profiles and clinical characteristics for the worsening of kidney function and for a rapid decline in kidney function. At the conclusion of this proposed work, the investigators will have an improved understanding of the natural history of CKD in sickle cell anemia. With the limited available therapies for the treatment of albuminuria in SCD and the paucity of data on the long-term efficacy of available pharmacotherapies, identification of biomarkers for the progression of CKD will facilitate the development of treatments which may be more effective than the current "standard of care."

ELIGIBILITY:
Inclusion Criteria:

1. age of 18 to 65 years;
2. confirmed diagnosis of sickle cell anemia (HbSS and SB0 thalassemia);
3. non-crisis, "steady state" with no severe pain episodes requiring medical contact during the preceding 4 weeks;
4. ability to understand the requirements of the study and be willing to give informed consent.

Exclusion Criteria:

1. bone marrow transplantation;
2. history of long-standing diabetes mellitus with suspicion for diabetic nephropathy as determined by a nephrologist;
3. known diagnosis of hepatitis B or C infection (patients will not be screened specifically for this during the study);
4. known HIV positive (patients will not be screened specifically for this);
5. history of cancer, except non-melanoma skin cancer;
6. pregnant or breastfeeding;
7. connective tissue disease such as SLE;
8. known glomerular disease unrelated to SCD;
9. patients with ESRD on chronic dialysis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HbSS or HbSB0 thalassemia between the ages of 18 and 65 years who meet the eligibility criteria and provide consent to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-11-17 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Age- and sex-adjusted rate of change, over 36 - 48 months, in estimated glomerular filtration rate in patients with sickle cell anemia | 36-48 months
  Estimated glomerular filtration rate will be ascertained using the CKD EPI equation
Age- and sex-adjusted rate of change, over 36 - 48 months, in albuminuria in patients with sickle cell anemia | 36-48 months
  Evaluate the rate of change in albuminuria by spot urine measurements of albumin-creatinine ratio during designated study visits
Cross-sectional association of biomarkers of endothelial function with kidney function (estimated glomerular filtration rate and albuminuria) in patients with sickle cell anemia | 36-48 months
  Plasma levels of ET-1, VEGF and soluble VCAM-1 from samples obtained at designated study visits will serve as measures of endothelial function
Cross-sectional association of urine and plasma metabolomics profiles with kidney function (estimated glomerular filtration rates and albuminuria) in patients with sickle cell anemia | 36-48 months
  Untargeted metabolic profiling of plasma and urine will be performed using high-resonance nuclear magnetic resonance spectrometry. Plasma and urine analytes which are significantly associated with estimated glomerular filtration rate and albumin-creatinine ratio will be ascertained.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Ataga, MD, Principal Investigator — UTHSC Center for Sickle Cell Disease
Locations (3):
- United States (3):
  - University of North Carolina-Chapel Hill, Chapel Hill, North Carolina
  - Ohio State Adult Sickle Cell Program, Columbus, Ohio
  - UTHSC Center for Sickle Cell Disease, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ataga KI, Brittain JE, Moore D, Jones SK, Hulkower B, Strayhorn D, Adam S, Redding-Lallinger R, Nachman P, Orringer EP. Urinary albumin excretion is associated with pulmonary hypertension in sickle cell disease: potential role of soluble fms-like tyrosine kinase-1. Eur J Haematol. 2010 Sep;85(3):257-63. doi: 10.1111/j.1600-0609.2010.01471.x. Epub 2010 Jun 3. PMID 20491879
- [Background] Ataga KI, Derebail VK, Archer DR. The glomerulopathy of sickle cell disease. Am J Hematol. 2014 Sep;89(9):907-14. doi: 10.1002/ajh.23762. Epub 2014 Jun 19. PMID 24840607
- [Background] Ataga KI, Brittain JE, Jones SK, May R, Delaney J, Strayhorn D, Desai P, Redding-Lallinger R, Key NS, Orringer EP. Association of soluble fms-like tyrosine kinase-1 with pulmonary hypertension and haemolysis in sickle cell disease. Br J Haematol. 2011 Feb;152(4):485-91. doi: 10.1111/j.1365-2141.2010.08410.x. Epub 2011 Jan 11. PMID 21223248
- [Derived] Zhou LY, Derebail VK, Desai PC, Elsherif L, Patillo KL, McCune P, Wichlan D, Landes K, Ogu UO, Nelson M, Loehr LR, Cronin RM, Tang Y, Cai J, Ataga KI. Persistent albuminuria and chronic kidney disease in adults with sickle cell anaemia: Results from a multicenter natural history study. Br J Haematol. 2024 Sep;205(3):1159-1169. doi: 10.1111/bjh.19636. Epub 2024 Jul 8. PMID 38978309